CLINICAL TRIAL: NCT04334603
Title: EXercise InTervention in Heart Failure (EXIT-HF): a Randomized Controlled Trial
Brief Title: EXercise InTervention in Heart Failure
Acronym: EXIT-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar do Porto (Other)
Collaborators: Universidade do Porto (Other); Aveiro University (Other)
Responsible Party: Principal Investigator, Mário André Silva Santos, Cardiologist, MD, PhD, Centro Hospitalar do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019.123
Record Dates: First submitted 2020-01-22; First posted 2020-04-06 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure
Keywords: Heart failure; Home-based exercise; Maximal oxygen consumption; Cost-effectiveness
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based exercise training (Experimental): The 12-week exercise-training program will include two sessions of combined exercise training per week, performed at home
  Interventions: Other: Exercise Training Program
- Clinical-based exercise training (Active Comparator): The 12-week exercise-training program will include two sessions of combined exercise training per week, performed at the hospital
  Interventions: Other: Exercise Training Program

INTERVENTIONS:
Other: Exercise Training Program — The 12-week exercise-training program will include two sessions of combined exercise training per week, performed at the hospital or at home.

SUMMARY:
This is a pragmatic, non-inferiority clinical trial, enrolling heart failure patients who will be randomized to a 12-week exercise training program either centre-based or home-based with telemonitoring. The impact of this intervention will be assessed on established surrogate markers in HF such as maximal exercise capacity, plasma biomarkers and quality of life. The cost-effectiveness and overall satisfaction with the treatment will also be studied. In addition to measure the clinical and economic impact of this innovative way of delivering exercise, it is intended to unravel new molecular pathways and assess a pool of biomarkers that provide a wide mechanistic picture underlying the clinical effects of exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HFrEF and HFpEF according to criteria of the European Society of Cardiology (2016)
2. Clinical stability for ≥ 6 weeks
3. Optimal medical treatment for ≥ 6 weeks
4. Patients that are able to understand and follow the exercise prescription
5. Written informed consent

Exclusion Criteria:

1. Patients who have undertaken cardiac rehabilitation within the past 12 months
2. Patients who have received an intracardiac defibrillator (ICD), Cardiac 3. Resynchronisation therapy (CRT) or combined CRT/ICD device implanted in the last 6 weeks
3. Inability to exercise or conditions that may interfere with exercise intervention
4. Signs of ischemia during cardiopulmonary exercise test
5. Comorbidity that may influence one-year prognosis
6. Symptomatic and/or exercise induced cardiac arrhythmia or conduction disturbances
7. Currently pregnant or intend to become pregnant in the next year
8. Expectation of receiving a cardiac transplant in the next 6 months
9. Participation in another clinical trial
10. Patients who are unable to understand the study information or unable to complete the outcome questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake (ml/kg/min) | Change from baseline in peak oxygen uptake (ml/kg/min) at 3 months
  Patients will be submitted to cardiopulmonary treadmill exercise tests at baseline and after 3 moths

SECONDARY OUTCOMES:
6-min walk test (6MWT) distance | Change from baseline to 3 months, and to 12 months.
  Changes in distance from the 6MWT.
Health status (EQ-5D-5L) | Change from baseline to 3 months, and to 12 months.
  Health status will be evaluated by the 5-level EQ-5D version (EQ-5D-5L) questionnaire. The questionnaire comprises five dimensions, each describing a different aspect of health (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has five response levels of severity which range from 0 (no problems) to 5 (extreme problems/ unable to do). In addition, there is a score of overall health range from 0 to 100%.
Health-related quality of life (MLHFQ) | Change from baseline to 3 months, and to 12 months.
  Health-related quality of life will be evaluated by the Minnesota Living with Heart Failure Questionnaire (MLHFQ). The MLHFQ is composed of 21 questions rated on a scale from 0 (no effect) to 5 (very much). The questionnaire is scored by summation of all 21 responses, where higher scores indicate worse quality of life.
Anxiety and Depression (HADS) | Change from baseline to 3 months, and to 12 months.
  Anxiety and Depression will be evaluated by the Hospital Anxiety and Depression Scale (HADS). The questionnaire is composed of 14 questions on a four-point (0-3) scale. The possible scores ranged from 0 to 21 for anxiety and 0 to 21 for depression. A score of 0 to 7 for either subscale will be regarded as being in the normal range, a score of 11 or higher indicating probable presence of the mood disorder and a score of 8 to 10 being just suggestive of the presence of the respective state.
Disutility | Evaluate at 3th month
  Individual disutility (inconvenience) perceived by patients and respective quality of life gains. Longevity to offset the exercise program disutility will be expressed in days.
Physical activity (steps/day) | Change from baseline to 3 months, and to 12 months.
  Physical activity will be assessed by a POLAR-M200 device with the numbers of daily steps.
Daily physical activity levels (min/day) | Change from baseline to 3 months, and to 12 months.
  Daily physical activity levels it will be measure with a POLAR-M200 device. Measures will be described as time spend in light physical activity, moderate and vigorous physical activity, and spend sitting or lying (minutes per day).
Dyspnea | Change from baseline to 3 months, and to 12 months.
  Dyspnea will be evaluated by the Dyspnea-12 (D-12) questionnaire. The D-12 consists of 12 descriptor items on a scale of none (0), mild (1), moderate (2), or severe (3). It provides an overall score for breathlessness severity that incorporates seven physical items and five affective items. Total scores from the D-12 range from 0 to 36, with higher scores corresponding to greater severity.
Mediterranean diet | Change from baseline to 3 months, and to 12 months.
  Adherence to Mediterranean diet will be evaluated by the 14-Item Mediterranean Diet Assessment Tool (MEDAS-14). The answer to each of the 14 items is scored with 1 in the case of meeting the criteria defined as typical of this type of food (range of possible variation 0-14 points). A total score ≥10 as represent a good adherence to the Mediterranean diet.
Hand grip strength | Change from baseline to to 3 and to 12 months.
  Hand grip strength will be assessed by Jamar dynamometer (kg)
Circulating number of endothelial progenitor cells, circulating endothelial cells, nitric oxide and endothelial Nitric Oxide Synthase | Change from baseline to 3 months
  These markers will inform endothelial function, damage and repair
Biomarkers (pg/ml) | Change from baseline to 3 months
  NTproBNP and ST2 (pg/ml)
Biomarkers (mg/L) | Change from baseline to 3 months
  hsCRP and Troponin (mg/L)
Concentration of plasma exosomes | Change from baseline to 3 months
  Plasma exosomes will be isolated using microbead-based sorting techniques and characterized by nanoparticle tracking analysis, Western blot, and quantitative real-time polymerase chain reaction assessments
Percentage of protein aggregates | Change from baseline to 3 months
  Protein aggregates (%) will be analysed using a diagonal two-dimensional (D2D) SDS-PAGE assay with mass spectrometry to identify and characterize detergent-resistant protein aggregates in plasma pre-cleared from albumin and immunoglobulin.
Cost-effectiveness of home-based exercise Vs. clinical-base exercise | At 12th month
  Compare cost effectiveness analysis of home-based exercise Vs. clinical-base exercise. The main outcome measure for this study will be cost per quality adjusted life year (QALY)
Physical fitness levels evaluation | Change from baseline to 3 and to 12 months.
  Physical fitness levels will be evaluated by the Senior Fitness test

OTHER OUTCOMES:
Exploratory analyses of urine proteome | Change from baseline to 3 months
  Exploratory analyses in urine protein will be performed to identify novel biomarkers predictive of exercise training therapeutic response. Urine of 10 patients from each group will be analyzed using a proteomic approach combining one-dimensional gel electrophoresis with liquid chromatography-tandem mass spectrometry (GeLC-MS/MS). Generated proteomic data will be analyzed with bioinformatic tools to reveal possible biomarkers of interest, that will be further validated by immuno-approaches such as ELISA or immunoblot.

CONTACTS AND LOCATIONS:
Overall Officials: Mário Santos, MD,PhD, Principal Investigator — Cardiology Service of Centro Hospitalar do Porto
Locations (1):
- Centro Hospitalar do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmidt C, Magalhaes S, Gois Basilio P, Santos C, Oliveira MI, Ferreira JP, Ribeiro F, Santos M. Center- vs Home-Based Cardiac Rehabilitation in Patients With Heart Failure: EXIT-HF Randomized Controlled Trial. JACC Heart Fail. 2025 May;13(5):695-706. doi: 10.1016/j.jchf.2024.09.024. Epub 2025 Jan 29. PMID 39895436